CLINICAL TRIAL: NCT00698347
Title: A Prospective, Non-controlled, Clinical Investigation of the M2a-Magnum™ Hip System
Brief Title: A Clinical Investigation of the M2a-Magnum™ Hip System
Status: Terminated | Type: Observational
Why Stopped: Centers would not continue follow-up; two centers transitioned patients to a new study.
Sponsor: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Other Study IDs: Biomet 12380-82
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis, Hip; Arthritis; Rheumatoid Arthritis; Joint Disease; Bone Disease
Keywords: Total Knee Replacement; Total Knee Arthroplasty; Hip Arthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis; Arthritis, Rheumatoid; Joint Diseases; Bone Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- M2a-Magnum™ Hip System: Patients who received the M2a-Magnum™ Hip System
  Interventions: Device: M2a-Magnum™ Hip System

INTERVENTIONS:
Device: M2a-Magnum™ Hip System
  Other Names: Magnum Hip

SUMMARY:
The purpose of this prospective clinical data collection is to document the performance and clinical outcomes of the M2a-Magnum™ Hip System

DETAILED DESCRIPTION:
This is a 10 year prospective data collection documenting the function and survivorship of the M2a-Magnum™ Hip System. Patients are required to come in for preoperative, operative, one year follow-up, three year follow-up, five year follow-up, and ten year follow-up exams.

This product was FDA cleared in 2004.

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory degenerative joint disease including: Avascular Necrosis, Diastrophic Variant, Fracture of the Pelvis, Fused Hip, Leg Perthes, Osteoarthritis, Slipped Capital Epiphysis, Subcapital Fractures, Traumatic Arthritis
* Rheumatoid Arthritis
* Correction of Functional Deformity
* Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques
* Revision of previously failed total hip arthroplasty

Exclusion Criteria:

Absolute contraindications include:

* Infection, Sepsis, and Osteomyelitis

Relative contraindications include:

* Uncooperative patient or patient with neurologic disorders that are incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, or neuromuscular disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that have already made the decision to undergo Total Hip Replacement and will receive the M2a-Magnum™ Hip System
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2004-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | 10 years

SECONDARY OUTCOMES:
Incidence of revisions, removals, and/or complications | Any time
X-Rays | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schenck, PhD, Study Director — Clinical Research, Biomet Orthopedics, LLC